CLINICAL TRIAL: NCT05692141
Title: The Value of Ultrasound Elastography for Differentiating Benign and Malignant Superficial Soft Tissue Masses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliaa Sayed Ali Hassan, Assuit, Assiut University
Other Study IDs: elastography
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Ultrasound Therapy; Complications
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound — For each lesion, ultrasound Elastography would be performed using a Linear probe ;

SUMMARY:
Ultrasonography has the advantages of being widely available, cost-effective, and allowing real-time dynamic examinations. Additionally, it is less time-consuming than magnetic resonance imaging (MRI) [1,2]. Recently developed ultrasound elastography techniques provide valuable information about intrinsic tissue properties by evaluating tissue elasticity, which may contribute to the diagnosis [3,4]. Ultrasound elastography can quantify and qualify tissue elasticity and add important information to the findings obtained by conventional ultrasonography [3,5-7]. Superficial soft tissue masses frequently occur and primarily manifest as benign lesions (including lipoma and hemangioma) that typically do not require treatment. Although malignant masses are rare, prompt surgical resections are required following the confirmation of a diagnosis (8). Therefore, differentiating between benign and malignant masses is important to prevent delays in the treatment of the malignant masses and avoid unnecessary surgical treatments for the benign masses (9). As the most effective method, pathological diagnosis is typically obtained from a needle biopsy. However, it is an invasive maneuver that is uncomfortable for patients and impractical for all types of soft tissue masses (10). Ultrasound is the primary examination method for superficial soft tissue masses to confirm their size, location, and the association between the masses and the surrounding structures. Through observations of the borders of the tissue masses, internal echo characteristics, and internal blood flow signals, ultrasounds may provide a preliminary diagnosis that is inaccurate (11). Stiffness of the tissue structures may be accessed using ultrasound elastography (UE) (12), which is an effective tool for differentiating malignant and benign masses (13). The stiffness of a malignant tumor is typically higher compared with a benign tumor. Previously, the differential diagnosis was primarily based on palpations by the physicians, which was indirect and could be limited in patients with obesity, mass sizes and depths, and physicians' experiences.

DETAILED DESCRIPTION:
The diagnostic imaging workup of soft tissue lesions begins with ultrasound and magnetic resonance imaging (MRI). In cases where the imaging features are not typical for a specific lesion (such as lipoma or ganglion cyst), imaging is insufficient to provide a definitive diagnosis, and these patients ultimately require a tissue sample by a percutaneous or excisional biopsy to guide further management.

In ultrasound, an emerging technology is an elastography which provides information on the stiffness of tissues. There are two main techniques, namely, strain elastography and shear wave elastography. In strain, or compression elastography, a force is applied to the tissues from the transducer by repetitive manual pressure, and the displacement (strain) is calculated from the return velocities of the tissues with respect to time. This creates a qualitative (color-coded) map of the elastic properties of the tissues. In shear wave elastography, vibration is applied to the tissues through a focussed ultrasound pulse, creating transverse shear waves in the tissues, the velocities of which can then be measured. Thus, shear wave elastography is a quantitative technique .

Patient selection This study will analyze patients who receive care at our institution patients with soft tissue masses. We retrospectively investigate patients' medical records, ultrasonographic exams, and histopathology reports Ultrasonographic Examination For each lesion, ultrasound Elastography would be performed using a Linear probe ; In Strain Elastography: Colors of the images represent different strain rates in decreasing order from red to green to blue. Based on the image colors, tissue elasticity was classified into 4 scores representing different stiffness: * score 1: completely red or green, * score 2: blue and green, with green as the dominant color, * score 3: blue and green, with blue as the dominant color, *score 4: completely blue. Strain rates of samples inside and outside the masses are measured to calculate the strain ratios (SRs).

In Shear Wave Elastography: The transducer is perpendicular to the lesion and stationary, without external compression. Grayscale images and color-coded histograms would be displayed with dual-mode imaging in real-time. In the chromatic scale, red indicates a higher shear modulus than blue. Several circular regions of interest (ROIs) with a diameter of 2 or 3 mm are placed within the lesion. The mean shear modulus for each ROI is measured automatically. We calculate the median value of several mean shear moduli corresponding to the ROIs, and this value is defined as the median shear modulus of the lesion. The unit of shear modulus values is the kilopascal (kPa)

ELIGIBILITY:
Inclusion Criteria:

* patients with superficial masses

Exclusion Criteria:

* inflammatory lesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will analyze patients who receive care at our institution patients with soft tissue masses. We retrospectively investigate patients' medical records, ultrasonographic exams, and histopathology reports
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
to investigate the value of ultrasound Elastography for differentiating benign and malignant superficial soft tissue masses . | baseline
  to investigate the value of ultrasound Elastography for differentiating benign and malignant superficial soft tissue masses .

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeoh HJ, Kim TY, Ryu JA. The feasibility of shear wave elastography for diagnosing superficial benign soft tissue masses. Ultrasonography. 2019 Jan;38(1):37-43. doi: 10.14366/usg.17059. Epub 2018 Jan 19. PMID 29580047